CLINICAL TRIAL: NCT05913661
Title: Prospective, Single-arm, Multicenter Phase II Study of Evaluation of the Efficacy and Safety of Pemigatinib Combined With PD-1 Inhibitor in First-line Treatment of Unresectable or Metastatic Intrahepatic Cholangiocarcinoma
Brief Title: Pemigatinib Combined With PD-1 Inhibitor in Unresectable or Metastatic Intrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: First Affiliated Hospital of Jinan University (Other); Shenzhen University General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-061-01
Record Dates: First submitted 2023-06-05; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-02

CONDITIONS: Carcinoma; Intrahepatic Cholangiocarcinoma; Digestive System Neoplasms; PD-1 Inhibitor; First-line Treatment
Keywords: unresectable intrahepatic cholangiocarcinoma; metastatic intrahepatic cholangiocarcinoma; first-line treatment; Pemigatinib; PD-1 inhibitor
MeSH Terms: conditions — Carcinoma; Cholangiocarcinoma; Digestive System Neoplasms | interventions — pemigatinib; Immune Checkpoint Inhibitors; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pemigatinib combined with PD-1 inhibitor (Experimental): pemigatinib combined with PD-1 inhibitor as first-line treatment within advanced unresectable or metastatic intrahepatic cholangiocarcinoma
  Interventions: Drug: Pemigatinib; Drug: PD-1 Inhibitors

INTERVENTIONS:
Drug: Pemigatinib — Pemigatinib is scheduled to be administered at a dose of 13.5 mg quaque die according to a 2-week dosing and 1-week discontinuation regimen.
  Other Names: Pemazyre
Drug: PD-1 Inhibitors — The dosing regimen is 200 mg IV Q3W
  Other Names: Sintilimab

SUMMARY:
This is a Prospective, single-arm, phase II study with multicenter participation. The objective of this study is to evaluate the efficacy and safety of pemigatinib combined with PD-1 inhibitor as first-line treatment for patients with advanced unresectable or metastatic intrahepatic cholangiocarcinoma.

DETAILED DESCRIPTION:
The study will be divided into two phases. The first phase is the safety import phase, in which three subjects with intrahepatic cholangiocarcinoma will be enrolled to receive a Scheduled dose of pemigatinib for one course of treatment， If the initial three subjects didn't develop DLT during the 21-day observation period, the dose will be considered tolerable and the study will proceed to Part II, otherwise, the dose will be adjusted and the evaluation will continue according to the above criteria.

A total of 30 subjects will be enrolled in Phase II of the study, and all screening-qualified subjects will receive pemigatinib combined with PD-1 inhibitor. pemigatinib and PD-1 inhibitors will be administered at established doses according to a regimen until progressive disease, intolerable toxicity, or informed consent form has been withdrawn. PD-1 inhibitors will be administered for a maximum of 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Local advanced, recurrent, or metastatic cholangiocarcinoma confirmed by histology or cytology and judged as unresectable by imaging and clinical diagnosis;
2. Have not received systematic treatment in the past;
3. The existence of FGFR2 fusion/rearrangement was confirmed by gene detection;
4. Male or female aged ≥ 18 years;
5. According to RECIST v1.1, there is at least one measurable target lesion. And the target lesion has not received local treatment;
6. No other anti-tumor treatment was received within 4 weeks before the first use of the study drug;
7. Life expectancy ≥ 12 weeks;
8. Eastern Oncology Collaboration group (ECOG) physical condition (PS) score 0-1;
9. Having sufficient organ and bone marrow function reserve, which is defined as follows:(1)Absolute neutrophil count (ANC) ≥ 1.5 × 109/L Platelet count (PLT) ≥ 80 × 109/L Hemoglobin content (HGB) ≥ 9.0 g/dL. G-CSF, GM-CSF, red blood cell infusion, and platelet infusion were not used within 14 days before the examination; (2)Liver function requirement for patients without liver metastasis: serum total bilirubin (TBIL) ≤ 1.5 × Upper limit of normal (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; Requirements for patients with liver metastasis or intrahepatic cholangiocarcinoma: serum TBIL ≤ 1.5 × ULN; ALT and AST ≤ 5 × ULN; (3)Renal function: creatinine clearance rate (Ccr) ≥ 50 mL/min (calculated by Cockcroft/Default formula): female: CrCl=(0.85 × (140 - Age) × (Weight)/(72 × Serum creatinine (mg/dL), male: CrCl=(140 age) × (Weight)/(72 × Serum creatinine (mg/dL); (4)Sufficient blood coagulation function, defined as the international standardized ratio (INR) or prothrombin time (PT) ≤ 1.5 times ULN; If the subject is receiving anticoagulation treatment, it is acceptable as long as PT is within the scope of anticoagulation drugs;
10. Female subjects of reproductive age or male subjects with female sexual partners of reproductive age shall take effective contraceptive measures during the whole treatment period and 6 months after the treatment period.

Exclusion Criteria:

1. Previously received selective FGFR inhibitor treatment, excluding pan target inhibitors such as Anlotinib and Lenvatinib
2. Received immunosuppressive drugs within 4 weeks before the first administration of the trial treatment, excluding local glucocorticoids or systemic glucocorticoids of physiological dose by nasal spray, inhalation, or other means (i.e. no more than 10 mg/day prednisone or other glucocorticoids of equivalent dose).
3. Received live attenuated vaccine within 4 weeks before the first administration of the trial treatment or during the study period.
4. Received any other study drug treatment or participated in interventional clinical research 4 weeks before the first administration of the trial treatment;
5. Before the first administration of the trial treatment, there was toxicity caused by previous anti-tumor treatment that was not restored to the level 0 or 1 of the National Cancer Institute Common Terminology Criteria for Adverse Events 5.0 (NCI CTCAE Version 5.0) (excluding alopecia, non-clinically significant laboratory abnormalities, and asymptomatic laboratory abnormalities).
6. Active, known or suspected autoimmune disease, or history of autoimmune disease in the past 2 years (patients with vitiligo that do not need systematic treatment, psoriasis, alopecia, or Graves' disease in the past 2 years, hypothyroidism who only need thyroid hormone replacement therapy and type I diabetes who only need insulin replacement therapy can be enrolled).
7. Known history of primary immunodeficiency.
8. Known to have active pulmonary tuberculosis.
9. Known Symptomatic central nervous system metastases and/or carcinomatous meningitis. For patients with brain metastasis who have received treatment in the past, if their condition is stable (no evidence of imaging progress is found at least 4 weeks before the first administration of the trial treatment), and repeated imaging examination proves that there is no evidence of new brain metastasis or enlargement of the original brain metastasis focus, and they do not need steroid treatment at least 14 days before the first administration of the trial treatment, they can participate in the trial. This exception does not include carcinomatous meningitis, regardless of its clinical stability should be excluded.
10. Medical history of other primary malignant tumors, except: (1)malignant tumors that have completely alleviated for at least 5 years before enrollment and do not require other treatment during the study period; (2)Fully treated non-melanoma skin cancer or malignant lentigo without evidence of disease recurrence; (3)Fully treated carcinoma in situ without evidence of disease recurrence.
11. During pregnancy or lactation.
12. Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
13. The following abnormal laboratory parameters: (1) Serum phosphate > ULN, and considered clinically significant by the investigator; (2) Serum calcium > ULN, or when serum albumin exceeds the normal range, the corrected calcium concentration of serum albumin exceeds the normal upper limit.
14. Known history of human immunodeficiency virus (HIV) infection or confirmed positive immune test result.
15. Known active serious infections or poorly clinically controlled infections.
16. Pleural fluid, ascites, or pericardial effusion with obvious clinical symptoms and requiring drainage.
17. Patients with acute or chronic active hepatitis B or hepatitis C, whose hepatitis B virus (HBV) DNA>2000 IU/ml or 10^4 copies/ml, or Hepatitis C virus (HCV) RNA>10^3 copies/ml, or Hepatitis B surface antigen (HBsAg) and anti HCV antibody were both positive. If laboratory parameters can be reduced to lower than the above standards after nucleotides antiviral treatment, the patient can be enrolled.
18. Clinically significant or uncontrolled heart diseases, including unstable angina, acute myocardial infarction within 6 months before the first administration of the trial treatment, New York Heart Association(NYHA) III/IV congestive heart failure, and uncontrolled arrhythmia (subjects with a pacemaker or atrial fibrillation with well-controlled heart rate can be enrolled).
19. There are ECG changes or medical history that the researchers consider clinically significant; For screening subjects with QTcF interval>480 ms and indoor conduction block (QRS interval>120 ms), JTc interval can be used to replace QTc interval after being approved by the sponsor (if so, JTc must be ≤ 340 ms).
20. Uncontrolled hypertension, systolic pressure>160 mmHg or diastolic pressure>100 mmHg after optimal medical treatment, hypertension crisis, or hypertensive encephalopathy history.
21. Hepatic encephalopathy, hepatorenal syndrome, or Child-Pugh B or more severe cirrhosis.
22. Patients with interstitial lung disease.
23. Major surgery (craniotomy, thoracotomy, or laparotomy) was performed within 4 weeks before the first administration of the trial treatment, or major surgery was expected to be performed during the study treatment.
24. Before starting treatment, the toxicity and/or complications of major surgery have not been fully recovered.
25. Pregnant or lactating females, or subjects who are expected to be pregnant or give birth during the study period from the screening follow-up to the completion of the safety follow-up (male subjects to 90 days after the last administration of the trial treatment).
26. Received radiotherapy within 4 weeks before the first administration of the trial treatment. The radiotherapy-related toxicity of the subject must have been fully recovered, and no corticosteroid treatment is required. It is confirmed that radiation pneumonia is excluded. For palliative radiotherapy for non-CNS diseases, a 2-week washout period is allowed.
27. History of disorder of calcium and phosphorus metabolism, or systemic electrolyte metabolism imbalance with ectopic calcification of soft tissues (excluding calcification of soft tissues such as skin, kidney, tendon, or blood vessel without systemic electrolyte metabolism imbalance caused by injury, disease, advanced age, and other reasons).
28. Corneal or retinal diseases with clinical significance confirmed by ophthalmological examination.
29. Received any potent CYP3A4 inhibitor or inducer was used 14 days or within 5 half-lives (whichever is shorter) before the first administration of the trial treatment. Ketoconazole is allowed for external use.
30. Known allergic reaction to pemigatinib or the excipients of the study drug pemigatinib.
31. Known hypersensitivity to any monoclonal antibody.
32. The investigator considered that the subject could not comply with the administration arrangement and study evaluation.
33. Unable to understand or unwilling to sign the Informed Consent Form (ICF).
34. Unable or unwilling to swallow pemigatinib or suffering from significant digestive system diseases that may interfere with absorption, metabolism, or excretion.
35. Known history of vitamin D deficiency and needed to supplement vitamin D beyond the physiological dosage (except for vitamin D dietary supplements).
36. Other acute or chronic diseases, mental diseases, or abnormal laboratory parameters that may lead to the following results: increase the risk related to the study participation or study drug administration, or interfere with the interpretation of the study results, and the patient is listed as ineligible to participate in the study according to the judgment of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-07 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 2 years
  The proportion of subjects who achieved complete response (CR; all target lesions disappeared) or partial response (PR; the sum of the longest diameter of target lesions decreased by ≥ 30%) according to the RECIST1.1 standard.

SECONDARY OUTCOMES:
Progression-Free-Survival | 2 years
  From the first administration to progressive disease[PD] or death.
Duration of Response | 2 years
  the period of time from the days which achieved complete response[CR] or partial response[PR] to progressive disease[PD]. This outcome measure is only applied to the subjects with objective remission
Disease Control Rate | 2 years
  The proportion of the sum of complete response[CR]、partial response[PR]、stable disease[SD] among the total cases.
Overall Survival | 2 years
  from the date of enrollment to Death

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, PHD, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Lei Zhang, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No